CLINICAL TRIAL: NCT00603109
Title: Effect of Rimonabant, a Cannabinoid Receptor 1 Antagonist on Weight Gain and Body Composition in Adults With Prader Willi Syndrome.
Brief Title: Effect of Rimonabant on Weight Gain and Body Composition in Adults With Prader Willi Syndrome
Acronym: PWS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Drug side effects leading to premature stop
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); PWSAUSA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0611008841
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2016-03

CONDITIONS: Prader-willi Syndrome
Keywords: Body weight, fat mass, growth hormone, ghrelin
MeSH Terms: conditions — Prader-Willi Syndrome; Body Weight | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Subjects receive rimonabant 20 mg per day PO
  Interventions: Drug: rimonabant
- II (Placebo Comparator): Subjects take placebo capsule one a day PO
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rimonabant — rimonabant capsule 20 mg per day PO for 6 months
  Other Names: Acomplia
  Arms: I
Drug: placebo — Subjects take 20 mg placebo capsule one a day PO for 6 months
  Arms: II

SUMMARY:
The purpose of this study is to evaluate the effect of rimonabant, a cannabinoid receptor-1 blocking drug, on the appetite, body weight, body fat and growth hormone level of subjects with Prader-Willi Syndrome (PWS). This will be a double blind placebo controlled clinical trial involving a total of 18 young adults aged 18 to 35 years with PWS. Patients will be divided in to the two groups of control and intervention, and treated with either placebo (inactive drug), or rimonabant 20 mg once a day for a total duration of 6 months. Body weight, fat distribution, objective and subjective assessment of the hunger, fasting blood sample for measurement of ghrelin and leptin (two hormones regulating appetite), serum lipids , IGF-1(growth hormone related protein), insulin and glucose concentrations will be measured upon enrollment, at 3 months, and at the end of the study. The proportion of body fat to muscle will be determined using a radiological technique, whole body dual-energy x-ray absorptiometry (DEXA) scan, and also by measurement of skin fold thickness, waist and hip circumference at the enrollment prior to the intervention, and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be selected if they have Prader Willi Syndrome previously confirmed by standard genetic testing (the DNA methylation test) or meet the clinical diagnostic criteria as follows :the presence of at least four of the six principal characteristics of PWS syndrome including 1) infantile hypotonia, 2) abnormal pubertal development, 3) obesity after early infancy, 4) dysfunctional central nervous system performance, 5) dysmorphic facial features, and 6) short stature. In addition, they must have one or more of the following characteristics commonly associated with PWS: 1) small hands and feet, 2) skin problems, 3) behavioral problems related to food, and 4) decreased pain sensitivity.
2. Subjects must be 18 to 35 years of age and fairly cooperative with the study protocol.
3. Subjects must have a BMI of at least 30 or more.

Exclusion Criteria:

1. Presence of pulmonary disease.
2. Presence of any other abnormal endocrine findings, including abnormal thyroid function.
3. Presence of significant behavioral problems or psychiatric illness including anxiety disorder and depression, interfering with the follow up of protocol. Any degree of depression and moderate to severe anxiety will be exclusion criteria for this study.
4. Subjects with Prader Willi Syndrome who are on other medications including growth hormone therapy, anti epileptic medications, or antipsychotic medications.
5. The presence of moderate to severe renal or liver disease. Mild elevations of liver enzymes are not exclusive.
6. Subjects who are on any other research or weight loss medication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Body Weight and Body fat mass | 6 months

SECONDARY OUTCOMES:
IGF-1, Leptin, Ghrelin, Serum Lipids and insulin sensitivity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roja Motaghedi, MD, Principal Investigator — NYPH-Weill Cornell Medical College; Moris Angulo, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- New York Presbyterian Hospital-Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deal CL, Tony M, Hoybye C, Allen DB, Tauber M, Christiansen JS; 2011 Growth Hormone in Prader-Willi Syndrome Clinical Care Guidelines Workshop Participants. GrowthHormone Research Society workshop summary: consensus guidelines for recombinant human growth hormone therapy in Prader-Willi syndrome. J Clin Endocrinol Metab. 2013 Jun;98(6):E1072-87. doi: 10.1210/jc.2012-3888. Epub 2013 Mar 29. PMID 23543664
- [Result] Motaghedi R, Lipman EG, Hogg JE, Christos PJ, Vogiatzi MG, Angulo MA. Psychiatric adverse effects of rimonobant in adults with Prader Willi syndrome. Eur J Med Genet. 2011 Jan-Feb;54(1):14-8. doi: 10.1016/j.ejmg.2010.09.015. Epub 2010 Oct 20. PMID 20965292